CLINICAL TRIAL: NCT02234414
Title: Pilot Study on the Epidemiology, Identification Rate and Treatment Penetration of Vertebral Fractures Due to Osteoporosis in Switzerland (SwOF)
Brief Title: Epidemiology, Identification Rate and Treatment Penetration of Osteoporotic Vertebral Fractures in Switzerland
Acronym: SwOF
Status: Completed | Type: Observational
Sponsor: Prof. Dr. med. Kurt Lippuner (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. med. Kurt Lippuner, President, Interessengemeinschaft Osteoporose
Organization: Interessengemeinschaft Osteoporose (Other)
Other Study IDs: IGO-SwOF 01
Record Dates: First submitted 2011-06-29; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Postmenopausal Osteoporosis; Spinal Fractures
Keywords: vertebral fracture assessment (vfa); vitamin D
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Spinal Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

SUMMARY:
In Switzerland, the prevalence of vertebral fractures in community- dwelling women is unknown and the published data from the Swiss hospitals statistics represent only the tip of the iceberg. In addition, the percentages of women correctly identified with vertebral fractures due to osteoporosis and the treatment rate of these women with a drug proven to reduce the risk of further fractures are unknown. Furthermore, it is not known whether the prevalence of vertebral fractures differs between urban and rural areas or between mountain areas and plain country, e.g. due to possible differences in sun exposure (vitamin D production) and/ or in physical activity and/ or dietary habits.

Clinical signs and symptoms leading to the suspicion of vertebral fracture(s) lack either sensitivity (wall-occiput distance) or specificity (rib-pelvis distance). Whether a combination of both would improve sensitivity and specificity is unknown.

The gold standard for the diagnosis of vertebral fracture relies on antero-posterior and lateral X-Rays of the thoracic and lumbar spine. Despite standardization of X-Ray readings, a retrospective study of hospitalized elderly patients has shown that as many as 50% of the radiographic reports failed to note the presence of moderate to severe vertebral fractures. In a primary care setting, fewer than 2% of the women received diagnoses of osteoporosis or vertebral fracture, although expected prevalence is 20% to 30% and appropriate drug treatment was offered to only 36% of the diagnosed patients.

The recent availability of software for vertebral fracture assessment (VFA) coupled to DXA measurements allows for the detection of vertebral deformities, which is critical for management of osteoporosis, as the existence of such deformities substantially increases the risk of subsequent fracture. Recently published results show that VFA allows the diagnosis of a vertebral fracture. The sensitivity of VFA for detection of vertebral fractures compared to expert radiologist reading of X-ray is excellent for grade 2 and 3 fractures, ranging between 90-94%.

DETAILED DESCRIPTION:
Examinations

* Community-dwelling women from a random sample (address lists may be chosen from public and/ or private providers)
* Aged 65-79 yrs
* Written informed consent

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling women from a random sample (address lists may be chosen from public and/ or private providers)
* Aged 65-79 yrs
* Written informed consent

Exclusion Criteria:

* Patients who underwent spine surgery
* Not willing or not able to sign informed consent
* In patients not willing or not able to participate, the reason for denial will be recorded for future evaluation.

Ages: 65 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will be based on a representative (age categories, urban vs. rural, plain vs. mountain) stratified random sample taken from the general population of women living in urban/ suburban and country/ mountain regions (stratified for n = one third each, based on city code) in the german speaking part of Switzerland.
Sampling Method: Probability Sample
Enrollment: 303 (Actual)
Dates: Start 2009-02; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of vertebral fractures in community dwelling Swiss women aged 65-79 years | at the only study visit

SECONDARY OUTCOMES:
Specificity, sensitivity, positive predictive value and negative predictive value for the prediction of underlying vertebral fracture of selected risk factors, clinical signs and vitamin D level, alone or in combination | at the only study visit
Assessment of the percentage of women correctly identified with a vertebral fracture and adequately treated for underlying osteoporosis and | at the only study visit
Assessment of the differences between these women and those who are either not correctly diagnosed or not correctly treated | at the only study visit

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Lippuner, Prof. Dr., Principal Investigator — Interessengemeinschaft Osteoporose
Locations (3):
- Switzerland (3):
  - Kantonsspital Olten, Olten
  - HFR Tafers, Tafers
  - Hochgebirgsklinik Davos, Wolfgang